CLINICAL TRIAL: NCT00535119
Title: A Phase 1 Study of ABT-888 in Combination With Carboplatin and Paclitaxel in Advanced Solid Malignancies
Brief Title: Veliparib, Carboplatin, and Paclitaxel in Treating Patients With Advanced Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00258; NCI-2009-00258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PCI-07-015; CDR0000566233; UPCI # 07-015 (Other: University of Pittsburgh Cancer Institute (UPCI)); 7967 (Other: CTEP); N01CM00038 (NIH); P30CA047904 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-04

CONDITIONS: Adult Solid Neoplasm; BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Hereditary Breast and Ovarian Cancer Syndrome
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Carboplatin; Paclitaxel; Taxes; veliparib

ARMS (1):
- Treatment (enzyme inhibitor therapy and chemotherapy) (Experimental): Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 3 and veliparib PO twice daily on days 1-7 until the recommended phase II dose is determined. Treatment repeats every 3 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial is studying the side effects and best dose of veliparib when given together with carboplatin and paclitaxel in treating patients with advanced solid cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving veliparib together with carboplatin and paclitaxel may help kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended dose for phase II studies of veliparib (ABT-888 ) that can be administered in combination with carboplatin and paclitaxel in patients with advanced solid malignancies. (Stratum I) II. To determine the recommended dose for phase II studies of veliparib that can be administered in combination with carboplatin and paclitaxel in patients with advanced solid malignancies that harbor a germline BRCA1/2 mutation. (Stratum II) (added 04/07/09)

SECONDARY OBJECTIVES:

I. To define the dose-limiting toxicity and other toxicities associated with the use of this combination.

II. To obtain preliminary evidence of antitumor activity in patients treated with this combination.

III. To evaluate the pharmacokinetic parameters of veliparib, carboplatin, and paclitaxel when administered as a combination.

IV. To conduct correlative science studies.

OUTLINE: This is a multicenter, dose-escalation study of veliparib. Patients are stratified according to BRCA status (no [stratum I] vs yes [stratum II]).

Patients receive carboplatin intravenously (IV) over 30 minutes and paclitaxel IV over 3 hours on day 3 and veliparib orally (PO) twice daily on days 1-7 until the recommended phase II dose is determined. Treatment repeats every 3 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo peripheral blood mononuclear cell collection periodically for pharmacokinetic and biomarker studies.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid malignancy
* Patients enrolled in stratum II of the study must have BRCA1/2 mutation (added 04/07/09)
* Patients with CNS metastases must be stable after therapy for CNS metastases (such as surgery, radiotherapy or stereotactic radiosurgery) for > 3 months and must be off steroid treatment prior to study enrollment
* ECOG performance status 0-2
* Life expectancy > 12 weeks
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 3 weeks since prior radiotherapy
* Prior veliparib allowed

Exclusion Criteria:

* Known history of allergic reactions to veliparib, carboplatin, or Cremophor-paclitaxel
* Uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Psychiatric illness or social situations that would preclude compliance with study requirements
* Peripheral neuropathy > grade 1
* Inability to take oral medications on a continuous basis
* Active seizure or history of seizure disorder
* Evidence of bleeding diathesis
* Received > 3 prior chemotherapy regimens for advanced stage disease for patients enrolled in stratum I (there is no upper limit on the number of prior regimens for patients enrolled in stratum II) (added 04/07/09)

  * Adjuvant chemotherapy administered ≥ 2 years prior to enrollment to the study does not count as a prior chemotherapy regimen
* Other concurrent investigational agents
* Concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) for each stratum | Up to 4 weeks
  The RP2D for each cohort will be defined by the study separately. Standard up & down dose-escalation scheme to determine the RP2D will be use, and toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) | During course 1
  Toxicities should be attributable to the study drug(s) to constitute DLT. Patients will be considered evaluable for DLT if they are eligible, and if they receive any amount of treatment and experience DLT or complete the first course of treatment
Frequency of platinum-DNA adducts | At baseline and 4 weeks post-treatment
  Changes will be summarized as means and standard deviations. A statistical test of the null hypothesis of no change in each variable will be done using the Wilcoxon signed-ranks procedure. Measurements of the two variables at additional time points will be analyzed in a descriptive fashion using tables and plots.
Incidence of stable disease (SD) | Measured from the start of the treatment until the criteria for progression are met, assessed up to 4 weeks post-treatment
  SD is defined as neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter (LD) since the treatment started.
PAR levels | Up to 4 weeks post-treatment
  Changes will be summarized as means and standard deviations. A statistical test of the null hypothesis of no change in each variable will be done using the Wilcoxon signed-ranks procedure. Measurements of the two variables at additional time points will be analyzed in a descriptive fashion using tables and plots.
Responses to veliparib in combination with carboplatin and paclitaxel | Up to 4 weeks post-treatment
  Response will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Time to progression (TTP) | Time from start of treatment to time of progression, assessed up to 4 weeks post-treatment
  Progression will be evaluated in this study using the new international criteria proposed by RECIST. TTP will be displayed for all patients and for patients who have responded; no formal statistical analysis is planned.
Toxicities as assessed by CTCAE v.4.0 | From the time of their first treatment with veliparib to up to 4 weeks post-treatment
  Toxicities will be defined as regimen-related if they are possibly, probably or definitely related to treatment. The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category, grade and dose level. Serious (≥ Grade 3) toxicities will be described on a patient-by-patient basis and will include any relevant baseline data.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, Principal Investigator — University of Pittsburgh Cancer Institute (UPCI)
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania